CLINICAL TRIAL: NCT04941248
Title: The Application of Total-body 13N-NH3 PET/CT to Study the Blood Perfusion System in the Whole Body
Brief Title: Total-body 13N-NH3 PET/CT to Study the Blood Perfusion in Whole Body
Status: Recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Yumei Chen, deputy head of the department of nuclear medicine, RenJi Hospital
Other Study IDs: KY2021-086
Record Dates: First submitted 2021-06-15; First posted 2021-06-28 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Cardiac Output
Keywords: Total-body; PET/CT; N-13 ammonia; Blood perfusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Healthy controls: All healthy subjects will undergo the following intervention: 13N-NH3 PET/CT scan on the total-body uEXPLORER scanner.
  Interventions: Device: total-body PET/CT(uEXPLORER , United Imaging Healthcare, China)
- Patients with decreased cardiac function: All patients will undergo the following intervention: 13N-NH3 PET/CT scan on the total-body uEXPLORER scanner.
  Interventions: Device: total-body PET/CT(uEXPLORER , United Imaging Healthcare, China)

INTERVENTIONS:
Device: total-body PET/CT(uEXPLORER , United Imaging Healthcare, China) — This prospective study will enroll twenty-five patients, including nine healthy volunteers, sixteen patients with decreased cardiac function . All of them will have a whole-body PET/CT(uEXPLORER , United Imaging Healthcare, China) in our department, Renji Hospital.

SUMMARY:
The aim of our study is to analyze and quantitate whole-body blood perfusion by total-body 13N-NH3 PET/CT(uEXPLORER), and evaluate the influence to other organs caused by the decreased cardiac function.

DETAILED DESCRIPTION:
Participants are invited to participate in a research that seeks to understand the dynamic blood perfusion in human body. The investigators expect to have twenty-five participants in this study at Renji Hospital, Shanghai. About sixteen of the participants will be patients who have been diagnosed with decreased cardiac function, nine participants will be healthy individuals with no known vascular disease. These healthy subjects will allow researchers to compare blood perfusion difference with those of persons with decreased cardiac function. All the participants will undergo the same procedure.

If participants agree to participate in this study, researchers will first interview participants and review the past medical record in order to document the medical history. When the screening procedures confirm that participants are eligible to participate in the study, participants will receive one dose of the non-therapeutic administration of a radioactive tracer called N-13 ammonia(13NH3) , then undergo one total body 13NH3 PET/CT Scan (uEXPLORER) to determine the blood flow value of the brain, kidney and other organs. The total body 13NH3 PET/CT Scan will allow investigators to observe and analyze the real-time blood flow differences between patients with between healthy controls and decreased cardiac function.

ELIGIBILITY:
Inclusion Criteria:

* Nine healthy volunteers with normal EF values
* Patients with decreased cardiac function, while their heart function grading above II(New York Heart Association,NYHA)
* Aged 60~90 years old
* Written informed consents will be offered and signed by all participants

Exclusion Criteria:

* History of vascular-related diseases in other organs
* Severe liver and kidney dysfunctions
* Patients who are pregnant or breast feeding
* People under the age of 60 years old
* Heart function grading below II(NYHA)
* inability to lie or to maintain posture in the scanner for one hour

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals aged between 60 and 90 years old with decreased cardiac function will be eligible for our enrollment; and participants without any history of vascular disease will be eligible.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2021-06-27 (Actual); Primary Completion 2025-12-08 (Estimated); Study Completion 2025-12-08 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Multi-Organ Blood Perfusion by Total Body Dynamic uEXPLORER PET/CT Scan | 4 years
  The total-body 13N-NH3 PET/CT will be adopted to evaluate the blood flow differences in whole body between healthy controls and patients with decreased cardiac function.

CONTACTS AND LOCATIONS:
Overall Officials: Yumei Chen, Ph.D; M.D., Principal Investigator — RenJi Hospital
Locations (1):
- Shanghai jiaotong University School of Medicine, Renji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benz DC, Ferro P, Safa N, Messerli M, von Felten E, Huang W, Patriki D, Giannopoulos AA, Fuchs TA, Grani C, Gebhard C, Pazhenkottil AP, Kaufmann PA, Buechel RR. Role of quantitative myocardial blood flow and 13N-ammonia washout for viability assessment in ischemic cardiomyopathy. J Nucl Cardiol. 2021 Feb;28(1):263-273. doi: 10.1007/s12350-019-01684-1. Epub 2019 Mar 20. PMID 30895563
- [Background] Lang JK, Canty JM Jr. The complexity of using resting myocardial perfusion to assess myocardial viability and predict functional recovery. J Nucl Cardiol. 2021 Feb;28(1):274-277. doi: 10.1007/s12350-019-01742-8. Epub 2019 May 13. No abstract available. PMID 31087267
- [Background] Kang KW, Kim JS, Cho SG, Kim J, Song HC. Acquisition of dynamic N-13 ammonia PET for myocardial blood flow quantification. J Nucl Cardiol. 2020 Aug;27(4):1288-1292. doi: 10.1007/s12350-020-02062-y. Epub 2020 Feb 19. No abstract available. PMID 32076961
- [Background] Giubbini R, Peli A, Milan E, Sciagra R, Camoni L, Albano D, Bertoli M, Bonacina M, Motta F, Statuto M, Rodella CA, De Agostini A, Calabretta R, Bertagna F; Italian Nuclear Cardiology Group (GICN). Comparison between the summed difference score and myocardial blood flow measured by 13N-ammonia. J Nucl Cardiol. 2018 Oct;25(5):1621-1628. doi: 10.1007/s12350-017-0789-z. Epub 2017 Feb 3. PMID 28160262
- [Background] Sciagra R, Lubberink M, Hyafil F, Saraste A, Slart RHJA, Agostini D, Nappi C, Georgoulias P, Bucerius J, Rischpler C, Verberne HJ; Cardiovascular Committee of the European Association of Nuclear Medicine (EANM). EANM procedural guidelines for PET/CT quantitative myocardial perfusion imaging. Eur J Nucl Med Mol Imaging. 2021 Apr;48(4):1040-1069. doi: 10.1007/s00259-020-05046-9. Epub 2020 Nov 2. PMID 33135093
- [Background] Lammertsma AA. Forward to the Past: The Case for Quantitative PET Imaging. J Nucl Med. 2017 Jul;58(7):1019-1024. doi: 10.2967/jnumed.116.188029. Epub 2017 May 18. PMID 28522743
- [Background] Akamatsu G, Uba K, Taniguchi T, Mitsumoto K, Narisue A, Tsutsui Y, Sasaki M. Impact of Time-of-Flight PET/CT with a Large Axial Field of View for Reducing Whole-Body Acquisition Time. J Nucl Med Technol. 2014 Jun;42(2):101-4. doi: 10.2967/jnmt.114.140665. Epub 2014 May 5. PMID 24799607
- [Background] Zhang X, Cherry SR, Xie Z, Shi H, Badawi RD, Qi J. Subsecond total-body imaging using ultrasensitive positron emission tomography. Proc Natl Acad Sci U S A. 2020 Feb 4;117(5):2265-2267. doi: 10.1073/pnas.1917379117. Epub 2020 Jan 21. PMID 31964808
- [Background] Zhang X, Xie Z, Berg E, Judenhofer MS, Liu W, Xu T, Ding Y, Lv Y, Dong Y, Deng Z, Tang S, Shi H, Hu P, Chen S, Bao J, Li H, Zhou J, Wang G, Cherry SR, Badawi RD, Qi J. Total-Body Dynamic Reconstruction and Parametric Imaging on the uEXPLORER. J Nucl Med. 2020 Feb;61(2):285-291. doi: 10.2967/jnumed.119.230565. Epub 2019 Jul 13. PMID 31302637
- [Background] Cherry SR, Jones T, Karp JS, Qi J, Moses WW, Badawi RD. Total-Body PET: Maximizing Sensitivity to Create New Opportunities for Clinical Research and Patient Care. J Nucl Med. 2018 Jan;59(1):3-12. doi: 10.2967/jnumed.116.184028. Epub 2017 Sep 21. PMID 28935835